CLINICAL TRIAL: NCT00889577
Title: Coronary Artery Disease and Its Association With Liver Steatosis Among HIV-Infected Persons
Status: Completed | Type: Observational
Sponsor: Henry M. Jackson Foundation for the Advancement of Military Medicine (Other)
Collaborators: Infectious Diseases Clinical Research Program (Other)
Responsible Party: Sponsor
Other Study IDs: IDCRP-018
Record Dates: First submitted 2009-04-28; First posted 2009-04-29 (Estimated); Last update posted 2023-03-21 (Actual); Status verified 2023-03

CONDITIONS: HIV Infections; Coronary Artery Disease; Non-Alcoholic Fatty Liver Disease
MeSH Terms: conditions — HIV Infections; Coronary Artery Disease; Non-alcoholic Fatty Liver Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Blood samples will be obtained
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The primary purpose of this study is to evaluate the association between nonalcoholic fatty liver disease (NAFLD) by computed tomography (CT) scan and coronary artery disease (CAD) measured by the calcium (CAC) score among HIV-infected persons.

ELIGIBILITY:
Inclusion Criteria:

* HIV patients who participated in our previous Liver Study, conducted at NMCSD, and HIV patients who did not participate in the Liver Study.

Exclusion Criteria:

* Women who are pregnant or breastfeeding will be excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: HIV positive patients who had participated in our previous Liver Study at NMCSD will be given the opportunity to participate in this study, as well as HIV patients who did not participate in the Liver Study.
Sampling Method: Non-Probability Sample
Enrollment: 233 (Actual)
Dates: Start 2008-12; Primary Completion 2010-03 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Coronary artery disease (CAD) measured by the CAC score | 1 year

SECONDARY OUTCOMES:
To determine the prevalence of coronary artery disease as determined by computed tomography (CT) of the coronary arteries among HIV patients, and to compare it to data from the general population using normative data from recent publications | 1 year
To evaluate predictors for coronary artery disease including demographics, concurrent conditions (e.g., diabetes, hyperlipidemia, tobacco use), and HIV factors such as ARV duration, HIV duration, and lipodystrophy | 1 year
To investigate the relationship between inflammatory markers (CRP, ESR), d-dimer, adiponectin levels, future inflammatory markers, and genetic polymorphisms with the presence of coronary disease and NAFLD | 1 year
To assess the relationship between increased pericardial fat on CT scan with visceral fat and cardiovascular disease | 1 year
To determine if Hounsfield units taken in the heart and aorta estimates hemoglobin levels | 1 year
To measure the pulmonary artery size to evaluate for prevalence of asymptomatic pulmonary hypertension among HIV-infected persons | 1 year
To describe the outcome of a positive CAC score in terms of follow-up test/procedure results to help describe the clinical significance of elevated scores. | 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- Naval Medical Center San Diego (NMCSD), San Diego, California, United States

REFERENCES:
- [Result] Norton L, Brodine SK, Medina S, Lemus H, Ricchiuti V, et al. (2013) Adiponectin Levels and Coronary Artery Disease among HIV-Infected Men. J AIDS Clin Res 4: 208.
- [Result] Crum-Cianflone N, Stepenosky J, Medina S, Wessman D, Krause D, Boswell G. Clinically significant incidental findings among human immunodeficiency virus-infected men during computed tomography for determination of coronary artery calcium. Am J Cardiol. 2011 Feb 15;107(4):633-7. doi: 10.1016/j.amjcard.2010.10.026. Epub 2010 Dec 31. PMID 21195379
- [Result] Medina S, Wessman D, Krause D, Stepenosky J, Boswell G, Crum-Cianflone N. Coronary aging in HIV-infected patients. Clin Infect Dis. 2010 Oct 15;51(8):990-3. doi: 10.1086/656442. No abstract available. PMID 20858081
- [Result] Crum-Cianflone N, Krause D, Wessman D, Medina S, Stepenosky J, Brandt C, Boswell G. Fatty liver disease is associated with underlying cardiovascular disease in HIV-infected persons(*). HIV Med. 2011 Sep;12(8):463-71. doi: 10.1111/j.1468-1293.2010.00904.x. Epub 2011 Jan 20. PMID 21251186
- [Result] Crum-Cianflone NF, Kathiria N, Shauger S, Love K, Boswell G. The association of epicardial adipose tissue with coronary artery calcification among HIV-infected men. AIDS. 2012 Jul 31;26(12):1573-6. doi: 10.1097/QAD.0b013e328355cef8. PMID 22713476